CLINICAL TRIAL: NCT02713048
Title: Sensitive Troponin I and Coronary Anatomy in Patients With Out-of-hospital Cardiac Arrest
Brief Title: Sensitive Troponin I in Out-of-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Marko Noc, Marko Noc, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: TnI OHCA
Record Dates: First submitted 2016-03-08; First posted 2016-03-18 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Arrest; Acute Coronary Lesion; Stable Obstructive Coronary Disease; Non-obstructive Coronary Disease
Keywords: Cardiac arrest; Troponin I; coronary anatomy
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acute coronary syndrome culprit coronary lesion
  Interventions: Other: Blood sample collection
- Stable obstructive coronary artery disease
  Interventions: Other: Blood sample collection
- Non-obstructive coronary artery disease
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Eight blood samples in each patient within 48 hours to perform Troponin I measurement.

SUMMARY:
Troponin is a major diagnostic criterion of acute myocardial infarction (AMI) which confirms myocardial damage and necrosis. In out-of-hospital cardiac arrest (OHCA) patients its dynamics and diagnostic value is often controversial and has not been well described. Most of prior studies were retrospective, using first generation troponin assays and assessing only admission troponin. The aim of this work is to correlate dynamics of sensitive troponin I with urgent coronary angiography.

Patients resuscitated after OHCA will be prospectively divided in three groups based on the results of their urgent angiographies. Serial assessment of sensitive troponin I will be obtained over initial 48 hours.

We expect admission troponin will not be predictive of AMI. Over next hours troponin levels will be highest in patients with acute coronary lesion, lower in stable obstructive coronary disease and insignificant in non-obstructive coronary disease. We also expect significant difference in highest values and dynamics of troponin in sub-group with spontaneous reperfusion (TIMI flow 2 and 3) comparing to patients with coronary occlusion (TIMI flow 0 and 1). In patients with non-obstructive disease we expect troponin levels to correlate with duration of cardiac arrest, number of external electric shocks and cumulative dose of adrenaline administered.

ELIGIBILITY:
Inclusion Criteria:

* female and male over 18 years old
* comatose survivors after out-of-hospital cardiac arrest (OHCA)
* absence of an obvious non-coronary cause
* urgent coronary angiography at admittance
* less than 3 hours from OHCA to first troponin assessment at admittance

Exclusion Criteria:

* sub-acute myocardial infarction
* coronary spasms or in-stent thrombosis within first 48 hours after admission
* Coronary surgery or death within first 48 hours after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose survivors after out-of-hospital cardiac arrest admitted to UMC Ljubljana
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2011-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Peak Troponin I value | Within 48 hours after hospital admission
  Peak troponin I values will be compared among 3 groups with different coronary anatomy

SECONDARY OUTCOMES:
Admission troponin I value | Within 3 hours of cardiac arrest
  Admission troponin I will be compared among 3 groups with different coronary anatomy
Peak troponin I value in acute coronary syndrome group | Within 48 hours after hospital admission
  Peak troponin I values will be compared among group with coronary artery occlusion and group with spontaneous reperfusion

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spaulding CM, Joly LM, Rosenberg A, Monchi M, Weber SN, Dhainaut JF, Carli P. Immediate coronary angiography in survivors of out-of-hospital cardiac arrest. N Engl J Med. 1997 Jun 5;336(23):1629-33. doi: 10.1056/NEJM199706053362302. PMID 9171064
- [Background] Dumas F, Cariou A, Manzo-Silberman S, Grimaldi D, Vivien B, Rosencher J, Empana JP, Carli P, Mira JP, Jouven X, Spaulding C. Immediate percutaneous coronary intervention is associated with better survival after out-of-hospital cardiac arrest: insights from the PROCAT (Parisian Region Out of hospital Cardiac ArresT) registry. Circ Cardiovasc Interv. 2010 Jun 1;3(3):200-7. doi: 10.1161/CIRCINTERVENTIONS.109.913665. Epub 2010 May 18. PMID 20484098
- [Background] Noc M, Fajadet J, Lassen JF, Kala P, MacCarthy P, Olivecrona GK, Windecker S, Spaulding C; European Association for Percutaneous Cardiovascular Interventions (EAPCI); Stent for Life (SFL) Group. Invasive coronary treatment strategies for out-of-hospital cardiac arrest: a consensus statement from the European association for percutaneous cardiovascular interventions (EAPCI)/stent for life (SFL) groups. EuroIntervention. 2014 May;10(1):31-7. doi: 10.4244/EIJV10I1A7. PMID 24832635
- [Background] Grubb NR, Fox KA, Cawood P. Resuscitation from out-of-hospital cardiac arrest: implications for cardiac enzyme estimation. Resuscitation. 1996 Nov;33(1):35-41. doi: 10.1016/s0300-9572(96)00971-9. PMID 8959771
- [Background] Mullner M, Oschatz E, Sterz F, Pirich C, Exner M, Schorkhuber W, Laggner AN, Hirschl MM. The influence of chest compressions and external defibrillation on the release of creatine kinase-MB and cardiac troponin T in patients resuscitated from out-of-hospital cardiac arrest. Resuscitation. 1998 Aug;38(2):99-105. doi: 10.1016/s0300-9572(98)00087-2. PMID 9863571
- [Background] Dumas F, Manzo-Silberman S, Fichet J, Mami Z, Zuber B, Vivien B, Chenevier-Gobeaux C, Varenne O, Empana JP, Pene F, Spaulding C, Cariou A. Can early cardiac troponin I measurement help to predict recent coronary occlusion in out-of-hospital cardiac arrest survivors? Crit Care Med. 2012 Jun;40(6):1777-84. doi: 10.1097/CCM.0b013e3182474d5e. PMID 22488008
- [Background] Voicu S, Sideris G, Deye N, Dillinger JG, Logeart D, Broche C, Vivien B, Brun PY, Capan DD, Manzo-Silberman S, Megarbane B, Baud FJ, Henry P. Role of cardiac troponin in the diagnosis of acute myocardial infarction in comatose patients resuscitated from out-of-hospital cardiac arrest. Resuscitation. 2012 Apr;83(4):452-8. doi: 10.1016/j.resuscitation.2011.10.008. Epub 2011 Oct 29. PMID 22037386
- [Background] Geri G, Mongardon N, Dumas F, Chenevier-Gobeaux C, Varenne O, Jouven X, Vivien B, Mira JP, Empana JP, Spaulding C, Cariou A. Diagnosis performance of high sensitivity troponin assay in out-of-hospital cardiac arrest patients. Int J Cardiol. 2013 Nov 30;169(6):449-54. doi: 10.1016/j.ijcard.2013.10.011. Epub 2013 Oct 16. PMID 24157232
- [Background] Keller T, Zeller T, Peetz D, Tzikas S, Roth A, Czyz E, Bickel C, Baldus S, Warnholtz A, Frohlich M, Sinning CR, Eleftheriadis MS, Wild PS, Schnabel RB, Lubos E, Jachmann N, Genth-Zotz S, Post F, Nicaud V, Tiret L, Lackner KJ, Munzel TF, Blankenberg S. Sensitive troponin I assay in early diagnosis of acute myocardial infarction. N Engl J Med. 2009 Aug 27;361(9):868-77. doi: 10.1056/NEJMoa0903515. PMID 19710485
- [Derived] Berden J, Steblovnik K, Noc M. Mechanism and extent of myocardial injury associated with out-of-hospital cardiac arrest. Resuscitation. 2019 May;138:1-7. doi: 10.1016/j.resuscitation.2019.02.026. Epub 2019 Feb 28. PMID 30826528